CLINICAL TRIAL: NCT03110354
Title: A Phase 1 Study of DS-3201b in Subjects With Acute Myelogenous Leukemia (AML) or Acute Lymphocytic Leukemia (ALL)
Brief Title: DS-3201b for Acute Myelogenous Leukemia (AML) or Acute Lymphocytic Leukemia (ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to slow accrual.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-A-U102
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Acute
Keywords: AML; ALL; Enhancer of zeste homolog (EZH) inhibitor; DS-3201b
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- DS-3201b 100 mg (Experimental): Participants who received 100 mg DS-3201b administered orally to participants with AML or ALL.
  Interventions: Drug: DS-3201b
- DS-3201b 150 mg (Experimental): Participants who received 150 mg DS-3201b administered orally to participants with AML or ALL.
  Interventions: Drug: DS-3201b
- DS-3201b 250 mg (Experimental): Participants who received 250 mg DS-3201b administered orally to participants with AML or ALL.
  Interventions: Drug: DS-3201b
- DS-3201b 500 mg (Experimental): Participants who received 500 mg DS-3201b administered orally to participants with AML or ALL.
  Interventions: Drug: DS-3201b
- DS-3201b 700 mg (Experimental): Participants who received 700 mg DS-3201b administered orally to participants with AML or ALL.
  Interventions: Drug: DS-3201b

INTERVENTIONS:
Drug: DS-3201b — DS-3201b is supplied as 25 and 100 mg capsules packaged in high-density polyethylene (HDPE) bottles.

SUMMARY:
This research study tests an investigational drug called DS-3201b. An investigational drug is a medication that is still being studied and has not yet been approved by the United States Food and Drug Administration (FDA). The FDA allows DS-3201b to be used only in research. It is not known if DS-3201b will work or not.

This study consists of two parts. The first part (Part 1) is a dose escalation that will enroll subjects with AML or ALL that did not respond or no longer respond to previous standard therapy. The purpose of Part 1 of this research study is to determine the highest dose a patient can tolerate or recommended dose of DS-3201b that can be given to subjects with AML or ALL. Once the highest tolerable dose is determined, additional subjects will be enrolled at that dose into Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Has AML or ALL and failed any prior induction therapy regimen or have relapsed after prior therapy
2. Has Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. Has adequate renal and hepatic function
4. Had at least 14 days for prior treatment to clear the body before initiation of DS-3201b administration (except for hydroxyurea that needs only 2 days for clearance)
5. Able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or comorbidity that would interfere with therapy.
6. Agrees to use an adequate method of contraception during the study and until 3 months after the last treatment.
7. Is willing to provide bone marrow biopsies and comply with protocol-defined evaluations
8. Has a life expectancy of at least 3 months

Exclusion Criteria:

1. Has presence of central nervous system (CNS) involvement of leukemia or a history of CNS leukemia
2. Has a second concurrent active primary malignancy such as solid tumor or lymphoma under active treatment
3. Has refractory nausea and vomiting, malabsorption, biliary shunt, significant bowel resection, graft versus- host disease (GVHD) significantly affecting gut motility or absorption, or any other condition that would preclude adequate absorption of DS- 3201b in the opinion of the treating physician and/or principal investigator (PI)
4. Has an uncontrolled infection requiring intravenous antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or tested positive for active hepatitis B or C infection
5. Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor
6. Has unresolved toxicities from previous anticancer therapy
7. Has received hematopoietic stem cell transplantation (HSCT) within 60 days of the first dose of DS-3201b
8. Has received concomitant treatment with a strong inhibitor or inducer of cytochrome P450 (CYP)3A4/5 within 7 days of first receipt of DS-3201b
9. Has consumed herbs/fruits that may have an influence on pharmacokinetics (PK) of DS-3201b from 3 days (14 days for St. John's wort) prior to the start of the study and throughout the entire study
10. Had major surgery within 4 weeks before study drug treatment
11. Has prolonged corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is > 450 milliseconds (ms) based on triplicate electrocardiograms (ECGs)
12. Is pregnant or breastfeeding
13. Has substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results
14. Has received prior treatment with enhancer of zeste homolog (EZH) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 participants who met all inclusion criteria and no exclusion criteria were enrolled in Part 1 of the study. Due to slow enrollment, Part 2 of the study or Dose Expansion was not conducted. No results are reported for Part 2.
Groups:
- DS-3201b 100mg: Participants who received 100 mg DS-3201b administered orally to participants with AML or ALL.
Period: Overall Study
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Started | 4 | 4 | 3 | 10 | 7
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 3 | 10 | 7
Not completed — Death | 1 | 0 | 0 | 1 | 0
Not completed — Start of new therapy | 0 | 0 | 0 | 0 | 1
Not completed — Failure to achieve response | 2 | 3 | 0 | 2 | 1
Not completed — Progressive disease | 1 | 1 | 3 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg | Total
Number analyzed (Participants) | 4 | 4 | 3 | 10 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 8 | 4 | 16
  >=65 years | 3 | 2 | 2 | 2 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (16.9) | 59.8 (27.7) | 64.7 (22.2) | 54.6 (16.0) | 55.9 (19.0) | 57.9 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 9 | 3 | 18
  Male | 2 | 2 | 1 | 1 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 3 | 7 | 5 | 22
  Black or African American | 0 | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade Treatment-emergent Adverse Event Classified as Dose-limiting Toxicities (Dose Escalation)
Description: Dose-limiting toxicity (DLT) is defined as a clinically significant non-hematologic treatment-emergent adverse event (TEAE) or abnormal clinical laboratory value that is clearly not related to disease progression, intercurrent illness, and occurring during the first cycle (28 days) on study that meets any of the following criteria: National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE), Version 4 Grade 3 aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), or bilirubin for ≥7 days; NCI-CTCAE Grade 4 AST (SGOT) or ALT (SGPT) of any duration; All Grade 4 non-hematologic toxicities of any duration; Any Grade 5 toxicity, unless proven to be clearly and incontrovertibly related to disease progression or intercurrent illness will constitute a DLT; All other clinically significant, non-hematological NCI-CTCAE Grade 3/4 AEs. AEs were coded using the MedDRA dictionary, Version 23.0.
Time Frame: Baseline up to Day 28
Population: Dose-limiting toxicities were assessed in the DLT Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 3 | 4 | 3 | 9 | 6
Participants
  Any TEAE classified as DLT, Any Grade | 0 | 0 | 0 | 1 | 3
  Gastrointestinal disorders, Any Grade | 0 | 0 | 0 | 0 | 2
  Diarrhea, Any Grade | 0 | 0 | 0 | 0 | 1
  Stomatitis, Any Grade | 0 | 0 | 0 | 0 | 1
  Blood and lymphatic system disorders, Any Grade | 0 | 0 | 0 | 0 | 1
  Bone marrow failure, Any Grade | 0 | 0 | 0 | 0 | 1
  Neoplasms benign, malignant, and unspecified (including cysts and polyps), Any Grade | 0 | 0 | 0 | 1 | 0
  Differentiation syndrome, Any Grade | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Who Experienced Any Grade Treatment-emergent Adverse Event (Dose Escalation)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug or has worsened after initiating the study drug until 30 days after the last dose of the study drug. AEs were coded using the MedDRA dictionary, Version 23.0.
Time Frame: Baseline up to 30 days after last study dose, up to approximately 4 years
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 4 | 4 | 3 | 10 | 7
Participants | 4 | 4 | 3 | 10 | 7

3. Secondary Outcome: Pharmacokinetic Parameter Maximum (Peak) Observed Concentration (Cmax) of DS-3201b
Description: Pharmacokinetic parameters were assessed using noncompartmental methods.
Time Frame: Cycle 1 Days 1 and 8 predose, 0.5, 1, 2, 4, 6, and 8 hours and Cycle 1 Day 15 postdose (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 4 | 4 | 3 | 10 | 7
ug/mL
  Cycle 1 Day 1 | 1.35 (0.98) | 1.09 (0.85) | 2.68 (1.06) | 3.82 (2.50) | 4.24 (2.30)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
  Cycle 1 Day 15 | 1.43 (1.80) | 0.73 (1.07) |  |  |
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 3 | 9 | 6
  Cycle 1 Day 8 |  |  | 3.69 (1.22) | 4.31 (1.84) | 5.31 (1.93)

4. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Observed Concentration (Tmax) of DS-3201b
Description: Blood samples were collected for PK analysis. PK parameters were assessed using noncompartmental methods.
Time Frame: Cycle 1 Days 1 and 8 predose, 0.5, 1, 2, 4, 6, and 8 hours and Cycle 1 Day 15 postdose (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 4 | 4 | 3 | 10 | 7
hours
  Cycle 1 Day 1 | 3.03 [2.00 to 4.25] | 4.06 [0 to 20.22] | 4.07 [2.17 to 4.18] | 3.81 [0 to 4.27] | 2.22 [1.02 to 8.00]
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 4 | 0 | 0 | 0
  Cycle 1 Day 15 | 2.00 [1.00 to 2.25] | 0 [0 to 2.08] |  |  |
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 3 | 9 | 6
  Cycle 1 Day 8 |  |  | 3.97 [2.03 to 4.00] | 4.03 [1.03 to 6.25] | 3.07 [0.68 to 7.97]

5. Secondary Outcome: Pharmacokinetic Parameter Area Under Plasma Concentration-Time Curve of DS-3201b
Description: Blood samples were collected for PK analysis. Area under the plasma concentration-time curve up to 24 hours (AUC24h) and area under the plasma concentration-time curve up to the last measurable concentration (AUClast) were assessed using noncompartmental methods.
Time Frame: Cycle 1 Days 1 and 8 predose, 0.5, 1, 2, 4, 6, and 8 hours and Cycle 1 Day 15 postdose (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 4 | 3 | 3 | 9 | 7
h*ug/mL
  Cycle 1 Day 1: AUC24h: number analyzed (Participants) | 2 | 1 | 3 | 9 | 5
  Cycle 1 Day 1: AUC24h | 8.97 (6.98) | 9.27 | 19.83 (4.71) | 43.13 (26.69) | 51.05 (26.55)
  Cycle 1 Day 15: AUC24h: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: AUC24h | 2.90 (1.71) |  |  |  |
  Cycle 1 Day 8: AUC24h: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4
  Cycle 1 Day 8: AUC24h |  |  |  | 46.34 (37.24) | 34.87 (2.36)
  Cycle 1 Day 1: AUClast | 7.79 (4.05) | 11.32 (7.62) | 19.79 (4.88) | 37.28 (23.64) | 41.58 (27.91)
  Cycle 1 Day 15: AUClast: number analyzed (Participants) | 4 | 1 | 0 | 0 | 0
  Cycle 1 Day 15: AUClast | 5.09 (6.01) | 8.23 |  |  |
  Cycle 1 Day 8: AUClast: number analyzed (Participants) | 0 | 0 | 3 | 9 | 6
  Cycle 1 Day 8: AUClast |  |  | 19.91 (4.85) | 20.75 (11.54) | 24.77 (11.70)

6. Secondary Outcome: Pharmacokinetic Parameter Trough Plasma Concentration (Ctrough) of DS-3201b
Description: Blood samples were collected for PK analysis. PK parameters were assessed using noncompartmental methods.
Time Frame: Cycle 1 Day 2 postdose (each cycle is 28 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
Number analyzed (Participants) | 4 | 4 | 3 | 9 | 7
ug/mL | 0.09 (0.05) | 0.58 (0.98) | 0.33 (0.11) | 0.64 (0.46) | 0.84 (0.76)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from baseline up to 30 days after last study dose, up to approximately 4 years.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug or has worsened after initiating the study drug until 30 days after the last dose of the study drug.
Arm/Group | DS-3201b 100mg | DS-3201b 150 mg | DS-3201b 250 mg | DS-3201b 500 mg | DS-3201b 700 mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/4 | 3/3 | 10/10 | 6/7
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 3/3 | 7/10 | 6/7
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 3/3 | 9/10 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-3201b 100mg (N=4) | DS-3201b 150 mg (N=4) | DS-3201b 250 mg (N=3) | DS-3201b 500 mg (N=10) | DS-3201b 700 mg (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2 | 2
Disease progression (General disorders) | 1 | 2 | 0 | 3 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-3201b 100mg (N=4) | DS-3201b 150 mg (N=4) | DS-3201b 250 mg (N=3) | DS-3201b 500 mg (N=10) | DS-3201b 700 mg (N=7)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear swelling (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Otorrhea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Extraocular muscle disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 2 | 4 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 4 | 4
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 3
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 2 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 2 | 1
Swelling face (General disorders) | 1 | 0 | 0 | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Stomatococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0
Coronavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Serum ferritim increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 1
Dysgeusia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 2
Headache (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03110354/Prot_SAP_000.pdf